CLINICAL TRIAL: NCT03690440
Title: OPTIBOT: Study Describing the Coverage, Cares and the Fertility of Patients of Less Than 45 Years With a Borderline Ovarian Tumor (BOT)
Brief Title: Study Describing the Coverage, Cares and the Fertility of Patients of Less Than 45 Years With a Borderline Ovarian Tumor
Acronym: OPTIBOT
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2017-09; N° : 2018-A00092-53 (Other: ID-RCB)
Record Dates: First submitted 2018-07-04; First posted 2018-10-01 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-03

CONDITIONS: Borderline Ovarian Tumors
Keywords: Borderline Ovarian Tumor (BOT); Fertility-sparing surgery; Gynecology; Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Retrospective and prospective multi-center study

Indication: Fertility-sparing surgery for patients with borderline ovarian tumor and fertility

Objectives:

* Description of the characteristics of the patients of less than 45 years having a fertility-sparing surgery for borderline ovarian tumors, the modalities of care and their fertility.
* Validation of a nomogram as an information medium to the patients concerned on their chance of alive birth according to their personal characteristics

Origin and nature of the specific data:

* Extraction from the database " Tumeurs Malignes Rares de l'Ovaire " (TMRO)
* Collection of retrospective further informations in the participating centers
* Data collection from the patients (questionnaires) The data will be identified by the TMRO number allocated to every participant of the TMRO study .

Data traffic :

TMRO database extraction for the patients with BOT and corresponding to the inclusion criteria, supplied by Arcagy-Gineco.

The database will be managed by the coordination team in an anonymous way by means of the patient identifiers of the TMRO base.

Enrichment of the base by the anonymous questionnaires filled by the patients and the complementary data transmissions of the centers on anonymised files.

ELIGIBILITY:
Inclusion Criteria:

* Women with history of Borderline Ovarian Tumor (BOT).
* Women who have had first a fertility-sparing surgery.
* Women old enough to procreate (= 45 years) during their first surgery.
* Women having agreed to participate in the previous study "Observatoire sur les Tumeurs Malignes Rares de l'Ovaire" (TMRO).
* Women who have not expressed their opposition to the research.

Exclusion Criteria:

* The patients who are not corresponding to the selection criteria are straightaway excluded from the retrospective database selected for the study (TMRO).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fertility-sparing surgery for patients with borderline ovarian tumor and fertility.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Description of the characteristics of the patients of less than 45 years having a fertility-sparing surgery for borderline ovarian tumors | December 2018
  Univariate and multivariate analysis on patients modalities of care and fertility , through medical history and questionnaires (study based on patients who were included in the previous study "Observatoire Sur Les Tumeurs Malignes Rares de l'Ovaire" (TMRO french network)

SECONDARY OUTCOMES:
Validation of a nomogram as an information medium to the patients concerned on their chance of alive birth according to their personal characteristics | December 2018
  Test of a published fertility prognostic tool in this population. Estimation of the precision of the estimation of alive birth in our cohort will be done by determining the difference between predicted live birth and observed rate of live birth.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine HEQUET, MD PhD, Study Director — Institut Curie
Locations (11):
- France (11):
  - Institut Bergonié, Bordeaux
  - Centre Jean PERRIN, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut Paoli CALMETTES, Marseille
  - Institut Curie, Paris, Paris
  - Hôpital Européen Goerges POMPIDOU, Paris
  - Goupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Centre Hospitalier Intercommunal Poissy - Saint-Germain, Poissy
  - Institut Curie - Saint-Cloud, Saint-Cloud
  - IUCT Oncopole - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine - Centre Alexis VAUTRIN, Vandœuvre-lès-Nancy